CLINICAL TRIAL: NCT06901609
Title: Effect of Genetic Polymorphism on the Clinical Outcome to SGLT2 Inhibitors in Heart Failure Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: National Heart Institute in Egypt (Unknown); Misr International University (Other); Princess Nourah bint Abdulrahman University, Riyadh, Saudi Arabia (Unknown)
Responsible Party: Principal Investigator, Neven Sarhan, Lecturer of Clinical Pharmacy, Misr International University
Other Study IDs: SGLT2 INHIBITORS
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure - NYHA II - IV; Cardiac Fibrosis; Cardiac Remodeling
Keywords: SGLT2 inhibitors; Heart Failure with reduced ejection fraction; Cardiac Remodeling
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected and stored in - 20°C environment for DNA extraction by DNA extraction kit according to manufacturer recommendation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort A: Newly diagnosed Heart Failure patients with reduced ejection fraction who are candidate for add-on treatment with sodium glucose transporter 2 inhibitor (SGLT2i) for the first time in addition to standard heart failure therapy.
  Interventions: Drug: SGLT2 inhibitor (Dapagliflozin 10mg)

INTERVENTIONS:
Drug: SGLT2 inhibitor (Dapagliflozin 10mg) — Renal response after 6 months of Dapagliflozin therapy among patients with heart failure reduced ejection fraction.

SUMMARY:
Heart failure with reduced ejection fraction (HFrEF) is a significant cause of morbidity and mortality. Sodium-glucose co-transporter-2 (SGLT2) inhibitors have demonstrated efficacy in improving renal outcomes in patients with HFrEF. Pharmacogenetics, the study of how genetic variations influence drug response, could elucidate inter-individual variability in treatment outcomes. This study aims to assess the impact of specific genetic variants on renal outcomes in HFrEF patients treated with SGLT2 inhibitors.

DETAILED DESCRIPTION:
Heart failure is broadly classified into two main types based on the left ventricular ejection fraction (LVEF): heart failure with preserved ejection fraction (HFpEF) and heart failure with reduced ejection fraction (HFrEF). HFpEF is characterized by a preserved or relatively normal LVEF, typically equal to or greater than 50%, despite signs and symptoms of heart failure. In contrast, HFrEF is defined by a reduced LVEF, typically less than or equal to 40%. [4] Accurate categorization of HF into HFpEF or HFrEF enables healthcare providers to implement targeted therapeutic approaches.

The intricate nature of heart failure necessitates a comprehensive approach to its diagnosis and management, given its varying presentations and underlying mechanisms. Heart injury, precipitated by diverse causes such as myocardial infarction, hypertension, and cardiomyopathies, triggers a complex and deleterious process of pathological remodeling and fibrosis within the cardiac tissue. This progressive cascade of events ultimately leads to the manifestation of heart failure. The pathophysiological mechanisms driving this progression are multifaceted, involving intricate cellular responses, neurohormonal activation, and inflammatory pathways. The initial insult, such as ischemic injury from myocardial infarction or chronic pressure overload from hypertension, sets in motion a series of maladaptive responses within the myocardium. These responses include cardiomyocyte hypertrophy, interstitial fibrosis, and alterations in extracellular matrix composition, which collectively impair myocardial contractility and promote ventricular dysfunction over time.

SGLT2 inhibitors, initially developed to manage blood glucose levels in patients with type 2 diabetes, now form part of the latest therapeutic strategies for heart failure as outlined in the 2022 AHA guidelines. This class, which includes empagliflozin, canagliflozin and dapagliflozin, has been shown to significantly reduce hospitalizations for heart failure and cardiovascular mortality in patients with symptomatic chronic HFrEF, irrespective of the presence of type 2 diabetes. Empagliflozin, a specific SGLT2I, has been particularly studied for its cardio-renal protective effects. Research by Miyata et al. (2021) has revealed that Empagliflozin goes beyond glycemic control by exerting beneficial effects on inflammatory and fibrotic markers.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with HFrEF (LVEF ≤40%).
* Initiation of SGLT2 inhibitor therapy.
* Stable background HF therapy for at least 4 weeks.
* Written informed consent for participation and genetic testing.

Exclusion Criteria:

* Known hypersensitivity to SGLT2 inhibitors.
* History of ketoacidosis or recurrent urinary tract infections.
* End-stage renal disease (eGFR <30 mL/min/1.73 m²).
* Life expectancy <6 months due to non-cardiovascular conditions.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure patients with reduced ejection fraction (LVEF<40%)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Reno-protective effect and gene polymorphism | 6 months
  Association between genetic polymorphism in SLC5A2, UMOD and ACE and Renal response in-terms of change in GFR among patients with heart failure.

SECONDARY OUTCOMES:
Gene polymorphisms and Renal biomarkers | 6 months
  Association between genetic polymorphism in SLC5A2, UMOD and ACE and Renal biomarkers among patients with heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem Zarif, MD, Study Chair — National Heart Institute
Locations (1):
- National Heart Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided